CLINICAL TRIAL: NCT03079037
Title: Circuit-Based Deep Brain Stimulation for Parkinson's Disease; Udall Project 1 Aim 2 and 3
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: NEUR-2016-22287
Record Dates: First submitted 2017-02-24; First posted 2017-03-14 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stimulation: Traditional deep brain stimulation
  Interventions: Device: Stimulation

INTERVENTIONS:
Device: Stimulation — Traditional deep brain stimulation

SUMMARY:
This study will test the hypothesis that deep brain stimulation (DBS) targeting specific changes in oscillatory activity at the site of stimulation will prove superior to continuous isochronal DBS thus providing the rationale for development and optimization of closed loop paradigms and determine whether the optimal closed-loop biomarker varies across subcortical targets, is task dependent, or serves to re-establish a default network that removes an underlying disruptive physiological state leading to greater improvement in motor signs and task performance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD
* DBS surgery or IPG battery replacement at UMN is planned as part of routine clinical care.

Exclusion Criteria:

* Other significant neurological disorder
* History of dementia
* Prior history of stereotactic neurosurgery
* Patients with post-operative complications or adverse effects (e.g. ON stimulation dystonias) that affect patient safety or confound the experiment will be excluded from further study
* Pregnant women

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's Disease (PD)
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2023-01-29 (Actual); Study Completion 2023-01-29 (Actual)

PRIMARY OUTCOMES:
Measure local field potential (LFP) changes in subthalamic nucleus (STN) and globus pallidus (GP) in OFF and ON states of stimulation and medication | 2 days
  Clinical ratings scales (MDS-UPDRS)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C. Park, MD/PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States